CLINICAL TRIAL: NCT04387760
Title: Treatment of Covid-19 With Favipiravir Versus Hydroxychloroquine: a Randomized Comparator Trial
Brief Title: Favipiravir vs Hydroxychloroquine vs Control in COVID -19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other)
Collaborators: Ebrahim Khalil Kanoo Community Medical Center (Unknown); Hereditary blood Disorder Centre - Salmaniya Medical Complex (Unknown); Mohammed Bin Khalifa Bin Sulman Al Khalifa Cardiac Centre, Awali (Unknown); Jidhafs COVID-19 Centre (Unknown); Sitra FICU (Unknown); Salmaniya Medical Complex- 6th Floor (Unknown); Salmaniya Medical Complex- Helipad (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40 / 07-May-2020
Record Dates: First submitted 2020-05-09; First posted 2020-05-14 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV 2; COVID-19
Keywords: Favipiravir; hydroxychloroquine; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; favipiravir

STUDY DESIGN:
Intervention Model Description: This is a parallel, prospective, interventional and randomized open label pilot trial involving 150 patients with COVID-19 disease. On confirmation of SARS-CoV-2 infection subjects will be randomised to hydroxychloroquine or favipiravir or standard clinical care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hydroxychloroquine (Experimental): Hydroxychloroquine is widely used to treat autoimmune diseases, due to its immunomodulatory properties, such as systemic lupus erythematosus and rheumatoid arthritis, with an excellent safety profile. In vitro studies have suggested that their mode of action in COVID-19 disease is blockade of SARS-CoV-2 transport from endosomes to endolysosomes, which appears to be a requirement to release the viral genome.
  Interventions: Drug: Hydroxychloroquine; Other: Routine care for COVID-19 patients
- Favipiravir (Experimental): Favipiravir is an antiviral drug that it is a pyrazinecarboxamide derivative with activity against influenza viruses, west nile virus, yellow fever virus, foot and mouth disease virus as well as against flaviviruses (i.e. arenaviruses, bunyaviruses and alphaviruses).
  Interventions: Drug: Favipiravir; Other: Routine care for COVID-19 patients
- Standard clinical care (Active Comparator): Supportive care according to local guidelines
  Interventions: Other: Routine care for COVID-19 patients

INTERVENTIONS:
Drug: Hydroxychloroquine — 400mg BID PO day 1 then 200mg BID PO from day 2 to day 10.
  In addition to Hydroxychloroquine all patients will receive the standard care (according to local Bahrain COVID19 guidelines). Any patient who is fit for discharge, can be discharged and medications will be stopped on discharge.
  Other Names: Hydroxychloroquine sulfate; Plaquenil
  Arms: Hydroxychloroquine
Drug: Favipiravir — 1600mg BID PO day 1600mg BID PO day 2 to day 10.
  In addition to Favipiravir all patients will receive the standard care (according to local Bahrain COVID19 guidelines). Any patient who is fit for discharge, can be discharged and medications will be stopped on discharge.
  Other Names: Avigan; T-705; favipira; favilavir
  Arms: Favipiravir
Other: Routine care for COVID-19 patients — Supportive care according to local guidelines
  Other Names: Standard clinical care

SUMMARY:
Hydroxychloroquine is widely used to treat autoimmune diseases. Clinical investigation has found that a high concentration of cytokines were detected in the plasma of critically ill patients infected with SARS-CoV-2, therefore, hydroxychloroquine as anti-inflammatory agents may reduce this response in accord with their use in autoimmune disease where the cytokine response can be reduced.

Favipiravir is an antiviral drug developed in Japan that the data sheet notes that it is a pyrazinecarboxamide derivative with activity against influenza viruses, west nile virus, yellow fever virus, foot and mouth disease virus as well as against flaviviruses, arenaviruses, bunyaviruses and alphaviruses. In February the drug was used for COVID-19 disease in China and was declared effective in treatment, and a report published (in press) comparing Favipiravir with Lopinavir /ritonavir suggested that Favipiravir was superior for prevention of disease progression and viral clearance.

The objective of this pilot study is to compare three arms: hydroxychloroquine; favipiravir; standard care (no specific SARS-CoV-2 treatment) only, in symptomatic patients infected by SARS-CoV-2 in an open label randomized clinical trial. The difference between groups will allow an effect size to be determined for a definitive clinical trial.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2/2019-nCoV) and has developed into a pandemic with serious global public health and economic sequelae. As of June 30, 2020 over 10,000,000 cases have been confirmed worldwide leading to over 500,000 deaths (https://coronavirus.jhu.edu/map.html). Currently no vaccine exists, however chloroquine and hydroxychloroquine have been documented as potentially having antiviral properties with efficacy against COVID-19 disease. Chloroquine is used in the treatment of malaria and amebiasis and is still used in the prophylaxis of malaria. Hydroxychloroquine sulfate is a derivative of Chloroquine that has been demonstrated to be much less (~40%) toxic than Chloroquine in animals. Hydroxychloroquine is widely used to treat autoimmune diseases, due to its immunomodulatory properties, such as systemic lupus erythematosus and rheumatoid arthritis, with an excellent safety profile. In vitro studies have suggested that their mode of action in COVID-19 disease is blockade of SARS-CoV-2 transport from endosomes to endolysosomes, which appears to be a requirement to release the viral genome. Clinical investigation has found that high concentrations of cytokines are detectable in the plasma of critically ill patients infected with SARS-CoV-2, suggesting that cytokine storm is associated with disease severity; therefore, Chloroquine/ hydroxychloroquine may reduce this response by acting as anti-inflammatory agents in accord with their use in autoimmune disease, where their reduction in cytokine response has been extensively researched and demonstrated.

Favipiravir is an antiviral drug developed in Japan (as noted in the data sheets) that it is a pyrazinecarboxamide derivative with activity against influenza viruses, west nile virus, yellow fever virus, foot and mouth disease virus as well as against flaviviruses (i.e. arenaviruses, bunyaviruses and alphaviruses). Its mode of action is through inhibition of viral RNA-dependent RNA polymerase. In February the drug was used for COVID-19 disease in China and was declared effective in treatment, and a report published (in press) comparing Favipiravir with Lopinavir /ritonavir suggested that Favipiravir was superior for prevention of disease progression and viral clearance.

"The Solidarity Trial" is a global pragmatic clinical trial being undertaken by WHO that aims to explore the efficacy of different treatment modalities for SARS-CoV-2. An application for Bahrain to join the study for collaboration has been made. In "The Solidarity Study" there will be four treatment modalities investigated, including chloroquine phosphate alone, remdesivir, lopinarvir with ritonavir or lopinarvir with ritonavir plus interferon. Favipiravir is not included, and therefore this study will not be replicating features of "The Solidarity Trial" but instead will provide additional and novel findings on favipiravir efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Admitted COVID-19 patients being treated as an in-patient at a hospital facility.
* COVID-19 diagnosis confirmed by PCR nasopharyngeal swab.
* Study participants must be symptomatic with any COVID-19 symptoms defined by the Bahrain National Protocol
* Onset of symptoms must be within 10 days prior to enrolment.
* Study participants must have the ability to give informed consent.
* Participants must be at minimum 21 years of age.
* Mild to Moderate COVID-19 disease defined as saturation equals to or more than 93% on room air or PaO2:FiO2 ratio more than 300 on enrolment.

Exclusion Criteria:

* Severe COVID-19 disease: defined as presence of SpO₂ less than 93% on room air or a PaO₂ to FiO₂ ratio of 300 or lower.
* Patients on ventilatory support.
* Cardiac dysfunction that would preclude treatment with hydroxychloroquine:

  1. Patients on medication known to prolong QT segment.
  2. Known history of LQT syndrome.
  3. Acquired QT prolongation at baseline >500ms.
  4. AV block.
  5. Bundle Branch Block.
  6. Known history of Cardiomyopathy, Pulmonary Hypertension, or Sick Sinus Syndrome.
  7. History of ventricular tachyarrhythmia.
  8. Patients with implantable cardioverter-defibrillator (ICD).
  9. Patients with a baseline bradycardia of less than 50 beats per minute.
* Renal dysfunction (estimated glomerular filtration rate less than 30ml/min).
* Hepatic dysfunction defined as:

  1. Transaminitis more than three times the upper limit of normal or
  2. Chronic liver disease of Child Pugh Class B or higher.
* Gout or a history of gout
* Patients that are pregnant or breastfeeding.
* Patients with a known allergy to an intervention medication.
* Patients who receive any of the study medications prior to randomization
* Patient with G6PD
* Readmission due to COVID19 disease.
* Participants in any other COVID-19 disease trial.
* Patients on immunosuppressants, HIV patients, cancer patients who received chemotherapy within the past 6 months, or who are on chronic oral steroids.
* Patients unable to give informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome is the Medial clinical scale at end of study follow up | Until discharge, death or for a maximum of 30 days or readmission
  Median clinical scale at end of study follow up (day 14 or on discharge/death, whichever is earlier)

SECONDARY OUTCOMES:
Requirement of Escalation of Respiratory Support | Until discharge, death or for a maximum of 14 days or readmission
  Implementation of escalation of Respiratory Support
Adverse effects(cardiac, renal, hepatic, hypoglycaemia (defined as RBS <3.9 mmol/L)) | Until discharge,death or for a maximum of 14 days or readmission
  Monitor and document all adverse effects during therapy
Requirement of ICU Admission | Until discharge, death or for a maximum of 14 days or readmission
  Deterioration of clinical condition requiring ICU admission
Mortality rate | Mortality will be collected up to 30 days
  30 days Mortality rate due to COVID-19
Readmission rate | Readmission will be collected up to 30 days from start of the study
  30 days readmission rate will be captured
Daily National Early Warning (NEWS) 2 Score | Until discharge, death or for a maximum of 14 days
  Daily NEWS 2 will be calculated which is a tool that improves the detection and response to clinical deterioration in adult patients and is a key element of patient safety and improving patient outcomes
Daily Sequential Organ Failure Assessment (SOFA) score | Until discharge, death or for a maximum of 14 days
  Daily SOFA score will be calculated which can identify the critical point at which patients exhibit the highest degree of organ dysfunction
Change in Laboratory indices | Until discharge, death or for a maximum of 14 days
  Determination of the change in D-dimer, ratio of Lymphocyte to Neutrophil, lactate before and after treatments as a measure of disease activity
Discharge and Length of Hospital Stay | Until discharge, death or for a maximum of 14 days
  Patients will be followed during their hospital stay until discharge
QT prolongation | Until discharge, death or for a maximum of 14 days or readmission
  Determination of the change in QT prolongation, before and after treatments as a measure of disease activity
Cardiac arrythmia (fatal and non fatal) | Until discharge, death or for a maximum of 14 days or readmission
  Detection of Cardiac arrythmia (fatal and non fatal), before and after treatments as a measure of disease activity
Viral clearance | until discharge, death or for a maximum of 30 days
  Viral clearance defined as a single negative SARS-CoV2 PCR nasopharyngeal swab

CONTACTS AND LOCATIONS:
Overall Officials: Manaf Al Qahtani, Dr., Principal Investigator — Royal College of Surgeons in Ireland - Bahrain
Locations (1):
- Royal College of Surgeons in Ireland - Bahrain, Manama, Bahrain

IPD SHARING:
Plan to Share IPD: Yes
Monitoring, audits, and REC review will be permitted and provide direct access to source data and documents. The Lead PI and the researchers assigned by him will have access to the stored data/specimens. Only the Lead PI and the researchers assigned working on this study will be eligible to obtain the data/specimens from the participants during data collection.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Dr Manaf will act as the data custodian and is responsible for the storage, handling and quality of the study data.
  Data will be collected in the case report form to allow for cross referencing to check validity.
  Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished. All essential documents including source documents will be retained for a period of 5 years after study completion (last patient, last study point). A label stating the date after which the documents can be destroyed will be placed on the inside front cover of the case notes of trial participants.
Access Criteria: Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished.

REFERENCES:
- [Background] McChesney EW. Animal toxicity and pharmacokinetics of hydroxychloroquine sulfate. Am J Med. 1983 Jul 18;75(1A):11-8. doi: 10.1016/0002-9343(83)91265-2. PMID 6408923
- [Background] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Delang L, Abdelnabi R, Neyts J. Favipiravir as a potential countermeasure against neglected and emerging RNA viruses. Antiviral Res. 2018 May;153:85-94. doi: 10.1016/j.antiviral.2018.03.003. Epub 2018 Mar 7. PMID 29524445
- [Background] Dong L, Hu S, Gao J. Discovering drugs to treat coronavirus disease 2019 (COVID-19). Drug Discov Ther. 2020;14(1):58-60. doi: 10.5582/ddt.2020.01012. PMID 32147628
- [Background] Cai Q, Yang M, Liu D, Chen J, Shu D, Xia J, Liao X, Gu Y, Cai Q, Yang Y, Shen C, Li X, Peng L, Huang D, Zhang J, Zhang S, Wang F, Liu J, Chen L, Chen S, Wang Z, Zhang Z, Cao R, Zhong W, Liu Y, Liu L. Experimental Treatment with Favipiravir for COVID-19: An Open-Label Control Study. Engineering (Beijing). 2020 Oct;6(10):1192-1198. doi: 10.1016/j.eng.2020.03.007. Epub 2020 Mar 18. PMID 32346491
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Birkett MA, Day SJ. Internal pilot studies for estimating sample size. Stat Med. 1994 Dec 15-30;13(23-24):2455-63. doi: 10.1002/sim.4780132309. PMID 7701146
- [Background] Senn SJ. Covariate imbalance and random allocation in clinical trials. Stat Med. 1989 Apr;8(4):467-75. doi: 10.1002/sim.4780080410. PMID 2727470
- [Background] Senn S. Testing for baseline balance in clinical trials. Stat Med. 1994 Sep 15;13(17):1715-26. doi: 10.1002/sim.4780131703. PMID 7997705
- [Background] Knol MJ, Groenwold RH, Grobbee DE. P-values in baseline tables of randomised controlled trials are inappropriate but still common in high impact journals. Eur J Prev Cardiol. 2012 Apr;19(2):231-2. doi: 10.1177/1741826711421688. No abstract available. PMID 22512015
- [Derived] AlQahtani M, Kumar N, Aljawder D, Abdulrahman A, Mohamed MW, Alnashaba F, Fayyad MA, Alshaikh F, Alsahaf F, Saeed S, Almahroos A, Abdulrahim Z, Otoom S, Atkin SL. Randomized controlled trial of favipiravir, hydroxychloroquine, and standard care in patients with mild/moderate COVID-19 disease. Sci Rep. 2022 Mar 23;12(1):4925. doi: 10.1038/s41598-022-08794-w. PMID 35322077